CLINICAL TRIAL: NCT01757730
Title: Magnetic Resonance Elastography as a Method to Estimate Stiffness of Soft Tissues
Acronym: MRE
Status: Recruiting | Type: Observational
Sponsor: Arunark Kolipaka (Other)
Responsible Party: Sponsor-Investigator, Arunark Kolipaka, Associate Professor, Ohio State University
Organization: Ohio State University (Other)
Other Study IDs: 2012H0027
Record Dates: First submitted 2012-12-18; First posted 2012-12-31 (Estimated); Last update posted 2025-04-06 (Actual); Status verified 2025-04

CONDITIONS: Heart Failure; Liver Fibrosis; Cardiac Transplant Rejection; Aortic Aneurysms
MeSH Terms: conditions — Heart Failure; Liver Cirrhosis; Aortic Aneurysm

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Altered Stiffness: Tissue stiffness will be evaluated in subjects those with disease conditions where stiffness changes from normal. These studies will be repeated for reproducibility.
- Healthy Volunteers: Tissue stiffness will be evaluated in normal subjects to determine the normal values. These studies will be repeated for reproducibility.

SUMMARY:
Magnetic resonance elastography is a novel non-invasive MRI technique to obtain stiffness of soft tissues such as liver, heart, kidneys, etc. In this imaging technique a person is laid in an MR scanner and a paddle (plastic drum) is put on the area of interest to send sound vibration via a speaker placed outside the scan room which is connecting plastic drum via a plastic tube. These vibrations are scanned using MRI to estimate the stiffness of soft tissues such as liver, heart, kidneys, breast etc.

DETAILED DESCRIPTION:
Recently a new and novel noninvasive imaging-based technique known as Magnetic Resonance Elastography (MRE) was developed that is capable of quantifying stiffness of soft tissues such as liver, spleen, kidney, heart brain, breast, aorta etc. In MRE a person is laid into an MR scanner which is similar to all MR scans. In addition, a drum (passive driver) is placed on the body (area close to the region of interest), which is connected by a long plastic tube that runs outside the scan room. This drum is tightly strapped by a Velcro to the body for better contact. Then the other end of the plastic tube is connected to an active driver that produces vibrations of frequencies in the range of 20Hz -2kHz. These frequencies of vibrations are transferred to the passive driver which produces vibrations on the body. These vibrations are tracked using MR scanner to produce wave images. A post-processing of these wave images are performed to obtain spatial stiffness maps. Currently, MRE is a clinical tool to assess hepatic fibrosis at many institutions. MRE is superior to many invasive techniques (i.e. biopsies, catheter based Pressure-Volume measurements) and mechanical testing in that it is noninvasive and can be performed in vivo under physiologic conditions. MRE could make stiffness widely available and could revolutionize the diagnosis and treatment of numerous diseases affecting stiffness of soft tissues. For example in Liver: diagnosis of hepatic fibrosis, Non-alcoholic fatty liver disease, liver tumors etc. Heart: diagnosis of diastolic dysfunction, myocardial infarction, hypertrophic cardiomyopathy, contractility etc. Aorta: Aortic aneurysms, hypertension etc. This technology is completely noninvasive and the vibrational energy is way below the required standards. Previous experiences of these vibrations are like massaging the body. The risks of this research study are minimal, which means that we do not believe that they will be any different than what you would experience at a routine clinical visit or during your daily life. This study will not make participants' health better. It is for the benefit of research.The specific aim of this study is that MRE can be used as a noninvasive tool to diagnose different disease states in soft tissues. In this study we will be applying this technique in adult volunteers to test the feasibility and validation of the technique in different organs.

ELIGIBILITY:
Inclusion Criteria:

Any participant 18 years or older and are MR safe.

Exclusion Criteria:

That study participants will be excluded if they have any unapproved metal in their bodies, or if the volunteers are pregnant or possible of becoming pregnant. Also if the participants are claustrophobic.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 1. You are 18 and over and affected by a certain disease condition such as Heart/Kidney/Lung/liver/spleen or aortic aneurysms or any other kind of diseases where stiffness of the soft tissue is thought to change.
  2. You are 18 and over and a healthy volunteer and not affected by any of the conditions mentioned in #1 above.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2012-03; Primary Completion 2028-03-01 (Estimated); Study Completion 2028-03-01 (Estimated)

PRIMARY OUTCOMES:
Stiffness of soft tissues | Participants will be followed for the duration of hospital stay, ecah clinical visit after discharge for an expected average up to 1 year
  Estimate any variation in stiffness

CONTACTS AND LOCATIONS:
Overall Officials: Arunark Kolipaka, PhD, Principal Investigator — Ohio State University
Locations (1):
- The Ohio State University Wexner Medical Center, Columbus, Ohio, United States

REFERENCES:
- [Result] Damughatla AR, Raterman B, Sharkey-Toppen T, Jin N, Simonetti OP, White RD, Kolipaka A. Quantification of aortic stiffness using MR elastography and its comparison to MRI-based pulse wave velocity. J Magn Reson Imaging. 2015 Jan;41(1):44-51. doi: 10.1002/jmri.24506. Epub 2013 Nov 15. PMID 24243654
- [Result] Chamarthi SK, Raterman B, Mazumder R, Michaels A, Oza VM, Hanje J, Bolster B, Jin N, White RD, Kolipaka A. Rapid acquisition technique for MR elastography of the liver. Magn Reson Imaging. 2014 Jul;32(6):679-83. doi: 10.1016/j.mri.2014.02.013. Epub 2014 Feb 13. PMID 24637083
- [Result] Kenyhercz WE, Raterman B, Illapani VS, Dowell J, Mo X, White RD, Kolipaka A. Quantification of aortic stiffness using magnetic resonance elastography: Measurement reproducibility, pulse wave velocity comparison, changes over cardiac cycle, and relationship with age. Magn Reson Med. 2016 May;75(5):1920-6. doi: 10.1002/mrm.25719. Epub 2015 Jun 12. PMID 26096227
- [Result] Wassenaar PA, Eleswarpu CN, Schroeder SA, Mo X, Raterman BD, White RD, Kolipaka A. Measuring age-dependent myocardial stiffness across the cardiac cycle using MR elastography: A reproducibility study. Magn Reson Med. 2016 Apr;75(4):1586-93. doi: 10.1002/mrm.25760. Epub 2015 May 22. PMID 26010456
- [Result] Moldovan L, Anghelina M, Kantor T, Jones D, Ramadan E, Xiang Y, Huang K, Kolipaka A, Malarkey W, Ghasemzadeh N, Mohler PJ, Quyyumi A, Moldovan NI. A module of human peripheral blood mononuclear cell transcriptional network containing primitive and differentiation markers is related to specific cardiovascular health variables. PLoS One. 2014 Apr 23;9(4):e95124. doi: 10.1371/journal.pone.0095124. eCollection 2014. PMID 24759906